CLINICAL TRIAL: NCT06149533
Title: A Randomized, Multicenter, Open-Label, Control, Clinical Trial to Evaluate the Efficacy and Safety of Edoxaban on Prevention of Catheter-related Thrombosis (CRT) in Cancer Patients
Brief Title: Evaluate the Efficacy and Safety of Edoxaban on Prevention of Catheter-related Thrombosis (CRT) in Cancer Patients
Acronym: Thrombosis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ma Fei，MD, Deputy Director of the Department of Medical Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCC4268
Record Dates: First submitted 2023-10-27; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Thrombosis, Venous; Cancer; Catheter Complications
Keywords: Prevention; Catheter-related Thrombosis; Cancer; Edoxaban
MeSH Terms: conditions — Venous Thrombosis; Neoplasms | interventions — edoxaban

STUDY DESIGN:
Intervention Model Description: A total of 366 patients with cancers who will be assessed as high risk by the thrombosis risk prediction model (refer to Appendix 1) are planned to be enrolled. All patients are planned to undergo anti-tumor chemotherapy and receive CVC or PICC catheterization on the first day of chemotherapy. The patients are randomly divided into the experimental group and the control group at a ratio of 1:1. The experimental group is treated with edoxaban to prevent catheter-related thrombosis, and the control group won't be treated with edoxaban.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The cohort 1 (Experimental): The cohort 1 is treated with edoxaban to prevent catheter-related thrombosis.
  Interventions: Drug: Edoxaban
- The cohort 2 (No Intervention): The cohort 2 won't be treated with edoxaban.

INTERVENTIONS:
Drug: Edoxaban — Edoxaban, an oral selective factor Xa inhibitor, had been approved by the National Medical Products Administration in 2018. It is used for the treatment and recurrence prevention of deep venous thrombosis (DVT) and pulmonary embolism (PE) in adults.
  Arms: The cohort 1

SUMMARY:
To evaluate the efficacy and safety of edoxaban in the prevention of tumor catheter-related thrombosis (CVC/PICC) in high-risk patients

DETAILED DESCRIPTION:
This study was a prospective, interventional, open, randomized controlled clinical study. A total of 366 patients with cancers who will be assessed as high risk by the thrombosis risk prediction model (refer to Appendix 1) are planned to be enrolled. All patients are planned to undergo anti-tumor chemotherapy and receive CVC or PICC catheterization on the first day of chemotherapy. The patients are randomly divided into the experimental group and the control group at a ratio of 1:1. The experimental group is treated with edoxaban to prevent catheter-related thrombosis, and the control group won't be treated with edoxaban. Venous vascular ultrasound will be conducted before the start of each cycle of chemotherapy or whenever patients have any thrombosis-related symptoms to assess whether they have catheter-related thrombosis. The incidence of catheter-related thrombosis during catheter. 1. The safety of edoxaban.2. The death caused by catheter-related thrombosis.3. The time of non thrombotic events.4. The incidence of venous thrombosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18.
2. Cancer patients with a catheter-related thrombus risk prediction model score ≥ 19.6.
3. ECOG score≤2.
4. Expected survival period over 6 months.
5. Malignant tumor was diagnosed by pathology and central venous catheterization was successfully completed.
6. Signing of informed consent voluntarily.

Exclusion Criteria:

1. Unknown location of the primary tumor.
2. Allergy to the active ingredient of edoxaban tablets or other excipients.
3. There is clinically significant active bleeding.
4. Platelet <50×109/L.
5. Liver disease with coagulopathy or clinically relevant bleeding risk.
6. A lesion or condition with a significant risk of major bleeding, such as current or recent gastrointestinal ulcer, recent brain or spinal injury, recent brain, spinal, or ophthalmic surgery, recent intracranial hemorrhage, esophageal varices, arteriovenous malformations, vascular aneurysms, or major intravertebral or intracerebral vascular malformations.
7. Concomitant therapy with any other anticoagulant, such as Unfractionated heparin (UFH), Low molecular heparin (Low molecular weight heparin, LMWH) (enoxaparin, dalteparin, etc.), heparin derivative (fondaparinux, etc.), oral anticoagulant (warfarin, dabigatran, rivaroxaban, apixaban, etc.), except in the special case of administration of UFH to maintain central venous catheter patency.
8. Surgical treatment is planned for the duration of the study.
9. Uncontrolled co-morbidities include, but are not limited to:

   Serious, uncontrolled infection. Symptomatic heart failure (New York Heart Association class II-IV) or symptomatic or poorly controlled arrhythmias Uncontrolled hypertension (systolic blood pressure ≥160mmHg or diastolic blood pressure ≥100mmHg) despite standard treatment.

   Any arterial thromboembolic event within 6 months before enrollment. Tumor invasion of large vessels. History of deep vein thrombosis, pulmonary embolism, or other major thromboembolism within 3 months before enrollment.
10. History of gastrointestinal perforation within 6 months before enrollment.
11. Pregnant or breastfeeding women.
12. Oral contraceptives.
13. Conditions considered unsuitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of catheter-related thrombosis during catheter | 6 months

SECONDARY OUTCOMES:
The incidence of bleeding caused by edoxaban | 6 months
  The incidence of bleeding caused by edoxaban including major bleeding, clinically relevant non-major bleeding and minor bleeding. The criteria is shown in Appendix 3.
The mortality rate caused by catheter-related thrombosis | 6 months
The time of non thrombotic events | 6 months
The incidence of venous thrombosis | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
These data involve patient privacy.